CLINICAL TRIAL: NCT06085937
Title: Feasibility and Safety of Single Dose Ketamine for Acutely Suicidal Patients in the Emergency Department
Brief Title: Feasibility and Safety of Ketamine for Suicidal Patients in the Emergency Department
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Lindsay Maguire, MD (Other)
Responsible Party: Sponsor-Investigator, Lindsay Maguire, MD, Assistant Professor of Emergency Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00150830
Record Dates: First submitted 2023-10-02; First posted 2023-10-17 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Suicide; Suicidal Ideation; Depression
MeSH Terms: conditions — Suicide; Suicidal Ideation; Depression | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ketamine (Experimental): All patients will receive the experimental drug.
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Patients will receive 0.2mg/kg of IV ketamine

SUMMARY:
There is currently no readily available pharmacologic intervention for suicidal ideation, a true psychiatric emergency, in the Emergency Department (ED). Investigators aim to trial low-dose, intravenous ketamine, a drug with well-established use in treatment-resistant depression, for patients who present to the ED with suicidal ideation.

DETAILED DESCRIPTION:
In this phase one trial, the investigators' objective is to establish the safety and feasibility of the study dose and route of administration, as well as to provide preliminary data on efficacy in reduction of depressive and suicidal symptoms as well as length of stay. Select patients will be given 0.2mg/kg of ketamine IV and observed in the ED for two hours. Vital signs and symptoms will be monitored. Patients will then be transferred to an admitting psychiatric hospital for definitive care as per standard of care. Surveys will be administered at times 0, 2 hours, 24 hours, and 72 hours to assess depressive and suicidal symptoms. ED providers and nursing staff will be asked to complete a short survey assessing ease of use and feasibility for ED administration for this purpose.

Specific aims are as follows:

1. To determine the safety of ketamine as a single IV dose in the ED for acutely suicidal patients.
2. To determine the feasibility of ketamine administration in the ED for the acutely suicidal patient.
3. To determine the impact of ketamine administration on depression and suicidal ideation in the acute phase as measured by the MADRS and C-SSRS.
4. To determine the impact on hospital length of stay calculated from ED arrival until discharge from admitting psychiatric hospital.

ELIGIBILITY:
Inclusion Criteria:

* Acutely Suicidality ("yes" answer to any of items 4 or 5 on C-SSRS "Suicidal Ideation" category)
* Require inpatient stabilization for SI or actions based on clinical observation and interview
* Are accepted for psychiatric stabilization at the University of Kansas Medical Center's Strawberry Hill campus
* Have a Glasgow Coma Score (GCS) of 15
* Age 18-65

Exclusion Criteria:

* Current or past history of psychosis
* Current or recent (past 4 weeks) symptoms of mania/hypomania as defined by Young Mania Rating Scale (YRMS) score of 12 or greater
* History of ketamine use disorder
* History of liver transplant
* Pregnancy or breastfeeding
* Imprisonment or inability to consent
* Positive urine drug screen or serum alcohol level
* Hypertension (SBP > 160 or DBP > 100 before administration of ketamine)
* Hypotension (SBP < 90)
* Presence of acute medical condition requiring admission to medical service
* Allergy, intolerance, or previous adverse reaction to ketamine
* Patient has 8+ lifetime ketamine exposures
* The treating physician determines that the patient is not a good candidate for the study (e.g. medical condition/procedure, medication that would contradindicate ketamine treatment)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | 2 hours
  Safety of use of ketamine for SI in the ED, as assessed by number and severity of reported serious adverse outcomes.
Provider and Nursing Attitudes toward use of Ketamine for Suicidal Patients in the ED [Feasibility] | 2 hours
  A questionnaire will be given to providers and nursing staff to assess [1] perceived safety, [2] provider comfort, [3] perceived efficacy, and [4] perceived feasibility for ED use as rated on a Likert scale from 1-5, with 5 relaying best perceived outcomes.

SECONDARY OUTCOMES:
Change in Suicidal Ideation | 72 hours
  Change of SI in ED patients after ketamine administration, as measured by the Columbia Suicide Severity Rating Scale (ideation subscore range 1-5, with higher number indicating increasing suicidal ideation; intensity subscore rating 2-25, with higher number indicating greater severity of suicidal ideation) and Montgomery-Asberg Depression Rating Scale.
Hospital Length of Stay | up to 2 weeks
  Impact of administration of ketamine on overall psychiatric hospital length of stay.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Kansas Strawberry Hill Campus, Kansas City, Kansas
  - University of Kansas Medical Center Emergency Department, Kansas City, Kansas